CLINICAL TRIAL: NCT03613779
Title: Efficacy of Lung Ultrasound Guided Therapy to Prevent Rehospitalizations in Heart Failure (CLUSTER-HF): a Randomized Controlled Trial
Brief Title: CLUSTER-HF: Lung Ultrasound Guided Therapy in Heart Failure
Acronym: CLUSTER-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Diego Araiza-Garaygordobil, Principal Investigator, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT-18-078
Record Dates: First submitted 2018-07-29; First posted 2018-08-03 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Heart Failure
Keywords: Lung ultrasound; Heart failure; Management
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LUS-guided therapy group (Experimental): LUS-guided therapy group. Patients randomly allocated to this arm will receive standard of care + LUS examination accessible to treating physician in every visit. Depending on the results of LUS examination, a low dose or high dose of diuretics will be administered.
  A standardized algorithm will be provided to ensure compliance to guideline-recommended medical therapy for heart failure.
  Interventions: Combination Product: LUS-guided therapy; Other: Standard of Care
- Control group. (Active Comparator): Control group. Patients randomly allocated to this arm will receive standard of care + LUS examination blinded to the treating physician in every visit. Diuretic titration will be based on standard practice (physical examination, symptoms and lab results).
  A standardized algorithm will be provided to ensure compliance to guideline-recommended medical therapy for heart failure.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Combination Product: LUS-guided therapy — Lung ultrasound guided therapy; if pulmonary congestion (more or equal than 3 B-lines), high dose (80-120mg PO/day furosemide) will be prescribed until next follow up re-assessment. If no congestion (less than 3 B-lines), low dose (0-40mg PO/day furosemide) will be prescribed until next follow up re-assessment
  Arms: LUS-guided therapy group
Other: Standard of Care — Standard of care will be provided.

SUMMARY:
Introduction: Heart failure is the leading cause of hospitalization among adults >65 years of age. Discharge from a heart failure hospitalization is followed by a 30 day readmission rate of ≈24%. Readmissions for heart failure are typically preceded by a gradual rise in ventricular filling pressures that begins days or weeks before any detectable changes in clinical status.

Lung ultrasound (LUS) is a tool that is easily available at bedside and shows superior sensitivity for the detection of pulmonary congestion when compared with X ray or physical examination, even in the absence of symptoms.

Pulmonary congestion assessed by LUS identifies a subgroup with worse prognosis and a higher rate of readmission and mortality. Whether the implementation of lung ultrasound in the follow up of heart failure patients may reduce the rate of readmissions is unknown.

Objective: The aim of this study is to evaluate a protocol of lung ultrasound guided therapy to prevent readmissions in heart failure outpatients.

Study design: the design of the investigator's study is a single center, single blinded, randomized controlled clinical trial.

Eligibility criteria: patients older than 18 years of age, who have been hospitalized for an acute heart failure syndrome. Exclusion criteria are life expectancy of less than 6 months, a surgically correctable cause of heart failure or uninterpretable lung ultrasound.

Eligible patients will be randomized into either "LUS-guided therapy group" or "control group" at hospital discharge. Follow-up visits will be scheduled at 15 days, 45 days, 3 months and 6 months after hospital discharge. LUS will be performed in all patients at hospital discharge and in every follow-up visit, but only in those allocated to the "LUS-guided therapy group" the information will be provided to the treating physician.

In the "LUS-guided therapy group", a prespecified diuretic dose will be administered to patients depending on the degree of ultrasonographic pulmonary congestion: if congestive (3 or more B lines, in total) a high dose (80-120mg furosemide PO/day) will be prescribed; if no congestive (less than 3 B lines, in total) a low dose (up to 40mg PO/day) will be prescribed.

Primary outcome will be the composite of hospital readmission + mortality. This study complies with the Declaration of Helsinki and the study protocol is being evaluated by the Ethic Committee of our institution.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the hospital with the primary or secondary diagnosis of heart failure
* The intra-hospital stay extends for at least 24 hours.
* The patient shows new symptoms (or worsening of known symptoms) due to the presentation of heart failure, including at least one of the following: dyspnea (dyspnea at rest, at exertion, orthopnea, nocturnal paroxysmal dyspnea), decreased exercise capacity, fatigue or other symptoms of target organ hypoperfusion or volume overload.
* The patient has at least two physical examination findings; or at least one finding to the physical examination and at least one complementary criterion, including: physical examination findings that are considered to be due to heart failure (peripheral edema, increase in the abdominal perimeter or ascites in the absence of primary liver disease, signs of pulmonary congestion including crackles, subcrepitant rales or decrease in vesicular murmur, increase in jugular venous pressure and / or hepatojugular reflux, gallop by third sound (S3) or rapid weight gain, clinically significant, attributed to water retention); and/or complementary findings that are considered to be due to heart failure, including Increase in levels of N-terminal-pro-BNP (NT-proBNP) compatible with decompensation of heart failure (> 2,000 pg / mL), radiographic evidence of pulmonary congestion, or invasive or non-invasive evidence of significant increase in ventricular filling pressures or decreased cardiac output.

Exclusion Criteria:

* Non interpretable lung ultrasound imaging or false positive findings (chronic lung interstitial disease, pneumonia, large pleural effusion).
* Lack of willing to provide informed consent
* Life expectancy lesser than 6 months
* Surgically correctable cause of heart failure (aortic stenosis, mitral regurgitation, multi-vessel coronary artery disease).
* Chronic kidney injury with an estimated or measured creatinine clearance rate lower than 15ml/min/1.73m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with the composite outcome of hospital readmission + mortality. | 6 months.
  Hospital readmission: urgent hospital non scheduled visit and stay of more than 24 hours, requiring medical interventions. Mortality: patient's death.
Number of patients with the composite outcome of hospital readmission + mortality + urgent visits for worsening HF | 6 months
  Hospital readmission: urgent hospital non scheduled visit and stay of more than 24 hours, requiring medical interventions. Mortality: patient's death. Urgent visits for worsening HF: non-scheduled visit to day care or ED that prompted increased oral / IV therapy, less than 24 hours stay.

SECONDARY OUTCOMES:
Quality of life measured by kansas city cardiomyopathy questionnaire (KCCQ) | 6 months
  Quality of life at 6 months assessed by KCCQ
NTproBNP concentrations | 6 months
  NTproBNP concentrations and change by last visit

CONTACTS AND LOCATIONS:
Overall Officials: Diego Araiza-Garaygordobil, MD, Principal Investigator — Instituto Nacional de Cardiología "Ignacio Chavez"
Locations (1):
- Instituto Nacional de Cardiología "Ignacio Chavez", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Second semester or 2020
Access Criteria: Via direct PI contact